CLINICAL TRIAL: NCT00005826
Title: Open Label Phase II Study on RFS 2000 (9-Nitro-Camptothecin, 9-NC) Administered as a "5 Days On-2 Days Off" Oral Treatment in Glioblastoma Multiforme
Brief Title: Nitrocamptothecin in Treating Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16996G; EORTC-16996G
Record Dates: First submitted 2000-06-02; First posted 2004-06-18 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — rubitecan

INTERVENTIONS:
Drug: rubitecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of nitrocamptothecin in treating patients who have glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the therapeutic activity and toxicities of nitrocamptothecin in patients with glioblastoma multiforme. II. Determine the overall response, duration of response, and progression free survival of these patients after this treatment.

OUTLINE: This is a multicenter study. Patients receive nitrocamptothecin orally daily on days 1-5. Treatment continues every 7 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 weeks until disease progression in the absence of further treatment.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed glioblastoma multiforme Recurrent disease confirmed by CT or MRI Bidimensionally measurable disease At least one lesion with the largest diameter at least 2 cm

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 times upper limit of normal (ULN) Alkaline phosphatase and transaminases no greater than 2.5 times ULN (no greater than 5 times ULN in case of liver metastases) Renal: Creatinine no greater than 1.7 mg/dL Cardiovascular: No history of ischemic heart disease in past 6 months Other: Not pregnant or nursing Fertile patients must use effective contraception No other prior or concurrent malignancies except cone biopsied carcinoma of the cervix or adequately treated basal or squamous cell skin carcinoma No other unstable systemic disease No active uncontrolled infection No psychological, familial, sociological, or geographical condition that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 6 weeks since prior adjuvant chemotherapy No other prior or concurrent chemotherapy allowed Endocrine therapy: Concurrent corticosteroids allowed Stable or decreasing dose for at least 2 weeks Radiotherapy: No high dose radiotherapy, stereotactic radiosurgery, or internal radiotherapy unless recurrence is histologically confirmed At least 3 months since prior radiotherapy to the brain Surgery: No prior surgery for recurrent brain tumor except biopsy At least 3 months since prior surgery for primary brain tumor Other: No other concurrent anticancer therapy No other concurrent investigational therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2000-03; Primary Completion 2000-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Raymond, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (13):
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- France (7):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lute Contre le Cancer,Georges-Francois Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Gustave Roussy, Villejuif
- Azienda Ospedaliera di Padova, Padua, Italy
- Academisch Ziekenhuis der Vrije Universiteit, Amsterdam, Netherlands
- Hospital Universitario 12 de Octubre, Madrid, Spain
- Switzerland (2):
  - Ospedale San Giovanni, Bellinzona
  - Clinique De Genolier, Genolier